CLINICAL TRIAL: NCT06709066
Title: Muscle Relaxant Effect and Safety of Mivacurium Chloride and Succinylcholine for Bronchoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peng Liang (Other)
Responsible Party: Sponsor-Investigator, Peng Liang, chief physician, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2024No.1625; ChiCTR (Registry Identifier: ChiCTR2400091276)
Record Dates: First submitted 2024-10-17; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia; Bronchoscopy; Muscle Relaxants
MeSH Terms: conditions — Muscle Hypotonia | interventions — Mivacurium; Succinylcholine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mivacurium chloride (Experimental): mivacurium chloride 0.14 mg/kg induction bolus + 0.5 mg/kg/h maintenance infusion
  Interventions: Drug: mivacurium chloride
- succinylcholine (Active Comparator): succinylcholine (1 mg/kg induction bolus + 5 mg/kg/h maintenance infusion)
  Interventions: Drug: succinylcholine

INTERVENTIONS:
Drug: mivacurium chloride — mivacurium chloride 0.14 mg/kg induction bolus + 0.5 mg/kg/h maintenance infusion
  Arms: mivacurium chloride
Drug: succinylcholine — succinylcholine (1 mg/kg induction bolus + 5 mg/kg/h maintenance infusion)
  Arms: succinylcholine

SUMMARY:
The goal of this clinical trial is to evaluate whether mivacurium chloride and succinylcholine can provide effective and safe muscle relaxation in adult patients aged 18-60 years undergoing bronchoscopy who require muscle relaxants during anesthesia. The main questions it aims to answer are:

* Is the recovery of spontaneous breathing within 15 minutes after drug discontinuation with mivacurium chloride non-inferior to succinylcholine?
* How do mivacurium chloride and succinylcholine compare in terms of intraoperative hemodynamics and post-operative recovery and comfort? Researchers will compare the mivacurium chloride group and the succinylcholine group to observe if mivacurium chloride can provide similar or better recovery effects compared to succinylcholine.

Participants will:

* Receive either mivacurium chloride (0.14 mg/kg induction bolus + 0.5 mg/kg/h maintenance infusion) or succinylcholine (1 mg/kg induction bolus + 5 mg/kg/h maintenance infusion) as a muscle relaxant during bronchoscopy.
* Have their vital signs, including blood pressure, oxygen saturation, and heart rate, monitored at multiple time points during the procedure.
* Be assessed post-procedure for spontaneous breathing recovery, consciousness recovery, and time to laryngeal mask airway (LMA) removal, as well as overall comfort and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for painless bronchoscopy who require muscle relaxants during anesthesia.
2. Aged between 18 and 60 years.
3. Classified as Grade I-III according to the American Society of Anesthesiologists (ASA) Physical Status Classification.
4. Patients voluntarily participate and sign an informed consent form.

Exclusion Criteria:

1. Patients with known allergies to any of the drugs involved in the study.
2. Patients with severe organic diseases of the brain, heart, lungs, liver, kidneys, or other major organs.
3. Patients with intracranial hypertension, asthma, cataracts, glaucoma, or other eye diseases.
4. Patients with myasthenia gravis, myasthenic syndrome, severe reduction or deficiency of cholinesterase, upper motor neuron injury, or upper motor neuron diseases that may cause abnormal responses to muscle relaxants.
5. Patients who have used medications affecting neuromuscular transmission function before the procedure.
6. Pregnant or breastfeeding patients.
7. Patients who have experienced extensive burns, acid-base imbalance, or electrolyte disturbances within the past six months.
8. Patients known or suspected to be homozygous for the atypical gene for plasma cholinesterase.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of spontaneous breathing recovery | Within 15 minutes after the completion of bronchoscopy.
  The rate of spontaneous breathing recovery after discontinuation of mivacurium chloride and succinylcholine during bronchoscopy.

SECONDARY OUTCOMES:
Recovery time of spontaneous breathing | From the end of bronchoscopy until spontaneous breathing, assessed up to 15 minutes post-procedure.
  Comparison of recovery times (minutes) for spontaneous breathing between mivacurium chloride and succinylcholine groups. Spontaneous breathing recovery is defined as achieving a tidal volume of 5 ml/kg and a respiratory rate of 12 breaths per minute.
Recovery time of consciousness | From the end of bronchoscopy until each specific recovery milestone is achieved, assessed up to 15 minutes post-procedure.
  Comparison of recovery times (minutes) for consciousness recovery. Consciousness recovery is defined as the ability to open eyes upon verbal command or when called by name.
Laryngeal mask airway (LMA) removal time | From the end of bronchoscopy until each specific recovery milestone is achieved, assessed up to 15 minutes post-procedure.
  Comparison of time to remove laryngeal mask airway (LMA) between mivacurium chloride and succinylcholine groups.
Mean pulse pressure at different stages | 3 minutes before induction, 1-minute intervals during induction until the LMA is inserted, 3 minutes after LMA insertion, 3 minutes after surgery start, 3 minutes after surgery end, and 3 minutes after LMA removal.
  Blood pressure measurements should be taken at 1-minute intervals during the induction phase (pre-LMA insertion), until the LMA is inserted. For the pre-induction phase, post-LMA insertion, surgery start, surgery end, and post-LMA removal, blood pressure should be measured every 3 minutes, with recordings taken for a total of 3 minutes at each stage. The average blood pressure (mmHg) for each stage was calculated using the values recorded during that stage for both the mivacurium chloride and succinylcholine groups.
Oxygen saturation (%) recorded at different stages | 3 minutes before induction, 1-minute intervals during induction until the LMA is inserted, 3 minutes after LMA insertion, 3 minutes after surgery start, 3 minutes after surgery end, and 3 minutes after LMA removal.
  Oxygen saturation (%) recorded for both mivacurium chloride and succinylcholine groups at different stages.
Heart rate recorded at different stages | 3 minutes before induction, 1-minute intervals during induction until the LMA is inserted, 3 minutes after LMA insertion, 3 minutes after surgery start, 3 minutes after surgery end, and 3 minutes after LMA removal.
  Heart rate recorded (beats per minute) at different stages for both mivacurium chloride and succinylcholine groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang X, Xu Y, Li J, Xi Y, Xu Z, Liang P. Effect and safety of mivacurium chloride and succinylcholine for bronchoscopy: study protocol for a single-center, randomized, non-inferiority, and positive-controlled clinical trial. Trials. 2026 Jan 22. doi: 10.1186/s13063-026-09463-3. Online ahead of print. PMID 41566470